CLINICAL TRIAL: NCT03431623
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of Subcutaneous CKD-11101 Versus Darbepoetin Alfa in Patients Who Had Renal Anemia Not on Dialysis
Brief Title: CKD-11101 Phase 3 SC Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136Ane14005
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multi-center, phase 3 clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-11101(Darbepoetin alfa) (Experimental): The dose of investigational product (Darbepoetin alfa) is adjusted according to the principles reflecting the MFDS (Ministry of Food and Drug Safety) approval for NESP, but is determined by the investigator's judgment considering various factors of the subjects that may affect the treatment of anemia.
  Interventions: Biological: CKD-11101(Darbepoetin alfa)
- NESP(Darbepoetin alfa) (Active Comparator): The dose of investigational product (Darbepoetin alfa) is adjusted according to the principles reflecting the MFDS (Ministry of Food and Drug Safety) approval for NESP, but is determined by the investigator's judgment considering various factors of the subjects that may affect the treatment of anemia.
  Interventions: Biological: NESP(Darbepoetin alfa)

INTERVENTIONS:
Biological: CKD-11101(Darbepoetin alfa)
  Arms: CKD-11101(Darbepoetin alfa)
Biological: NESP(Darbepoetin alfa)
  Arms: NESP(Darbepoetin alfa)

SUMMARY:
The aim of this study was to compare and evaluate efficacy and safety of subcutaneous CKD-11101 versus Darbepoetin alfa in patients who have renal anemia not on dialysis.

DETAILED DESCRIPTION:
This was designed as randomized, double-blind, multi-center, Phase 3 clinical study to evaluate the efficacy and safety of subcutaneous CKD-11101 versus Darbepoetin Alfa in patients who had stage 3, stage 4, and stage 5 chronic renal failure not on hemodialysis or peritoneal dialysis.

The selection criteria will be evaluated in patients who are receiving anemia correction among patients with 19 years of age or older and who had anemia in chronic renal failure of stage 3 or above.

Subjects who are identified to meet all inclusion criteria will be randomized to test group and control group at 1:1 ratio and go through 24-week correction period and efficacy evaluation period. During correction period and efficacy evaluation period, subjects will visit the clinical study center every 2 weeks to receive processes designated for each visit and be administered investigational product from the investigator in charge of drug administration.

In the safety evaluation period, all subjects will be administered test drug for 28weeks.

ELIGIBILITY:
* Inclusion Criteria

  1. Patients with 19 years of age or older
  2. Patients with chronic renal failure of stage 3 or above who are not on dialysis
  3. Patients with the Hb levels of 8 to 10g/dl measured at screening
  4. Patients with enough body iron stores who meet the following item:

     -Serum ferritin ≥ 100ng/ml or Transferrin saturation ≥ 20%
  5. Patients who have provided written consent to participate in the clinical trial voluntarily
* Exclusion Criteria

  1. Patients who are expected to need dialysis within a year or patients with rapidly progressive chronic renal failure
  2. Patients who have received drug treatment such as erythropoiesis stimulating agent for the purpose of correcting anemia within 12 weeks prior to screening
  3. Patients who have received red blood cell transfusion within 12 weeks prior to screening
  4. Patients with uncontrolled hypertension
  5. Patients who had hypersensitivity to erythropoietin agents
  6. Patients who had known hypersensitivity to mammalian cell-derived products or additives
  7. Patients with history of severe cardiovascular diseases
  8. Patients whose anemia is not caused by chronic renal failure or may affect anemia correction including the following conditions:
  9. Patients whose AST/ALT test results performed at screening exceeds twice of normal upper limit
  10. Patients who have experience of positive result in anti-erythropoietin antibody in previous treatment with erythropoiesis stimulating agent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changed amount of mean hemoglobin level in evaluation period compared to the baseline | ([Mean of hemoglobin measured in Weeks 20 - 24] - [Hemoglobin measured at Week 0])
  The equivalence test on mean hemoglobin level of test drug and reference drug administration groups in evaluation period (Weeks 20 - 24) compared to the baseline (Week 0) will be conducted.
Mean administration dose in evaluation period: Mean dose administered in Weeks 20 - 24 | Weeks 20 - 24
  The equivalence test on mean administration dose of test drug and reference drug administration groups in evaluation period (Weeks 20 - 24) will be conducted.

SECONDARY OUTCOMES:
Ratio of subjects who achieve target level of hemoglobin | Weeks 20 - 24
  Ratio of subjects who achieve target level of hemoglobin: Compare the number of subjects who achieve target level of hemoglobin during the evaluation period between groups
Days taken to reach target level of hemoglobin | Days taken to reach up to 24 weeks
  Days taken to achieve target level of hemoglobin: Compare days taken to achieve target level of hemoglobin between groups
Mean hemoglobin level for each week | Weeks 4, 8, 12, 16, 20, 24, and 52
  Mean hemoglobin level for each week: Compare Weeks 4, 8, 12, 16, 20, 24, and 52 between groups
Changed amount of mean hemoglobin level at Weeks 20, 24, and 52 compared to the baseline | Weeks 20, 24, and 52
  Compare the mean change of hemoglobin level at Weeks 20, 24, and 52 compared to the baseline
Ratio of subjects who receive transfusion | Weeks 0 - 24
  Ratio of subjects who receive red blood cell transfusion: Compare ratio of subjects who receive red blood cell transfusion during treatment period and evaluation period between groups

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Yang, M.D., Ph.D., Principal Investigator — yangch@catholic.ac.kr

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Lee JH, Ha Chung B, Joo KW, Shin SK, Kim YL, Na KY, Do JY, Park SK, Shin BC, Lee JS, Kim YW, Kim SW, Lee KW, Kang GW, An WS, Shin GT, Han S, Yang CW. Efficacy and safety of CKD-11101 (darbepoetin-alfa proposed biosimilar) compared with NESP in anaemic chronic kidney disease patients not on dialysis. Curr Med Res Opin. 2019 Jun;35(6):1111-1118. doi: 10.1080/03007995.2018.1560134. Epub 2019 Jan 17. PMID 30569763